# INFORMED CONSENT FOR TEACHERS AND EDUCATORS PARTICIPATING IN THE STUDY

The purpose of this document is to invite you to participate in the study entitled "Participatory Construction and Feasibility of a Multicomponent Intervention to improve the Well-being of Basic Education Children after the COVID-19 Pandemic", whose main investigator is Dr. Eva Madrid Aris , in conjunction with the co - investigators; Fanny Leyton Alvarez , Marcelo Briceño Araya, Karla Álvarez Kozubová , Carolina Godoy Peña, n, sponsored by the University of Valparaíso, for the development of the health research and development project – FONIS 2021.

So that you can make an informed decision, we will explain the procedures involved in carrying out the research, as well as what your collaboration would consist of:

1. This research will be carried out in Public Educational Establishments (EEP) with basic education in 2 sectors of Valparaíso, Mena and Reina Isabel II, during the year 2023.

# 2. Relevance of the study and benefits:

Child mental health is the foundation on which mental, physical and social health is built in adult life, prevention and early intervention of the problems investigated in this evolutionary stage is essential. Chile has a high prevalence of MS problems in childhood and adolescence. The school system is a privileged instance for the investigation of the emotional and behavioral problems of children and adolescents (NNA), but it has not always had a coordinated and functional intersectoral network to respond to the required demand. Therefore, this project seeks to contribute to the mental health of children and the school community through a multicomponent intervention. This program is based on a biopsychosocial mental health perspective that goes beyond the mere absence of disease, relieving protective resources, mainly those related to social support and networks necessary for human well-being. Therefore, the present research and interventions of the project aim to improve and install skills in basic education teachers, to early identify mental health difficulties that may occur in children with whom they maintain a daily relationship based on the teaching work, helping to generate timely and relevant access to the mental health programs of the territorial health network of the schools that will participate in the project, thanks to the articulation of intersectoral networks that will be promoted.

# 3. Objective:

The team of researchers hopes to know the real possibilities of the application and effectiveness, of an intervention that contemplates training teachers in the area of mental health in a hybrid modality, through a program co -constructed with the teachers participating in this research, in order to enhance their research capacities and referral to the public system of Chilean health, to promote access to a timely and relevant intervention, with the support of a network of institutions, from different sectors,

including; education, health, national service for minors, justice, neighborhoods among others.

# 4. Participation:

Your participation in this research is completely voluntary and you will not receive any payment for your agreement to participate. If you agree to participate, you must participate in a child mental health (SMI) literacy program, which will be carried out in a hybrid format (face-to-face and e-learning) and, if required, the application of the qualities and difficulties questionnaire (SDQ) that assesses emotional symptoms of the students you are in charge of, responding to an online questionnaire before and after the intervention on SMI and other mental health questionnaires, in addition, you may be asked for in-depth interviews to learn about your experience regarding the problems and facilitators that you identify in the implementation of the intervention.

## 5. Risks:

We make it clear that there are no potential risks in this study, neither physical, nor emotional, nor of any kind. On the other hand, the results would make it possible to have an intervention to improve SMI in EEP boys and girls, with its initial evidence on effectiveness and feasibility indicators, for its possible scaling up to the national level. Therefore, a study that has a favorable risk/benefit balance is considered.

# 6. Costs and payments:

If you agree to participate in the research project, you will not receive money as a payment for participation in the study. However, the participant declares to have the technological means of internet access to participate in the different activities described in this consent.

## 7. Rights of the participant:

By participating in this study, you have the right to express your doubts to the researcher at any time by email to <a href="mailto:eva.madrid@uv.cl">eva.madrid@uv.cl</a>. In addition, you can withdraw from the study at any time if you consider it necessary by communicating it to Dr. Eva Madrid, principal investigator; It should be noted that your withdrawal will not harm you in any way.

# 8. Confidentiality of the participant's identity

For the purpose of analysis and maintenance of databases, during the research process, all information related to names, places or other data that could later lead to the identification of the participants will be modified from the written and virtual records, instead it will be used a numeric code.

## 9. Confidentiality of data

The lists of information obtained from the participants will be maintained by the principal investigator in physical locations separate from the transcripts and the

audio and video recordings. While the transcriptions and audio and video recordings will be stored in a password-protected computer, which will be in a locked place and accessible only to researchers and therapists who participate in the processes. The protocol for the data protection chain will be explicitly established, which together with the informed consents will be stored in a safe place, to which only the researchers in charge of the project will have access. The criteria of the Singapore Declaration on Research Integrity will be taken into account. The project will take into account the criteria and recommendations of CONICYT and the Institutional Ethics Committee of the University of Valparaíso. All the transcripts of the committee meetings and focus groups will be made by the researchers, who will also participate in the data analysis process.

# 10. Use and Publication of the findings

The results of this study will be disseminated through different public channels, either in the form of publications (scientific articles) or presentations (exhibition in conferences and congresses). In addition, we hope that the technology that we will evaluate through this research will be transferred to public services later.

## 11. Evaluation of the Bioethics Committee and contact:

This research has been evaluated and accepted by the Institutional Committee of Bioethics of

Research in Human Beings from the University of Valparaíso. If you require it, you can contact any of its members with its administrative secretary, Ms. Patricia Arancibia Pardo, on the phone +56 32-2507909, or through the institutional email <a href="mailto:cec.uv@uv.cl">cec.uv@uv.cl</a>.

## 12. If you agree to participate, you will receive a copy of this document.

If the results of the instruments that measure health have a score of suspicion of mental health, you will be informed via mail or phone call and if you wish, this information will be delivered to the biopsychosocial team of the health network

| Name: | Researcher name: Eva Madrid Aris |
|-------|----------------------------------|
| RUT: | Investigator RUT: 6.890.922-8 |

Date: Date: Firm: Firm:

#### INFORMED CONSENT FOR GUARDIANS OF STUDENTS

The purpose of this document is to invite you to participate in the study entitled "Participatory Construction and Feasibility of a Multicomponent Intervention to improve the Well-being of Basic Education Children after the COVID-19 Pandemic", whose main investigator is Dr. Eva Madrid Aris, in addition to the following co - investigators; Fanny Leyton Alvarez, Marcelo Briceño Araya, Karla Álvarez Kozubová and Carolina Godoy Peña, sponsored by the University of Valparaíso, for the development of the health research and development project — FONIS SA21I0143 2021.

So that you can make an informed decision, the procedures involved in the execution of the investigation are detailed, as well as what your collaboration would consist of:

# 1. Research territory:

This research will be carried out in Public Educational Establishments (EEP) with basic education in 2 sectors of Valparaíso, Mena and Reina Isabel II, during the year 2023.

## 2. Relevance of the study:

Children's mental health is the foundation on which mental health (SM), physical and social in adult life is built; prevention and early intervention of the problems investigated in this evolutionary stage is essential. Chile has a high prevalence of MS problems in childhood and adolescence. The school system is a privileged instance for the investigation of the emotional and behavioral problems of children and adolescents (NNA). Therefore, this project seeks to contribute to the mental health of children and the school community through a multicomponent intervention. This research and interventions of the project aim to **improve and install skills in basic education teachers**, to early identify SM difficulties that may arise in children with whom they maintain a daily relationship based on teaching work, **contributing to generate a timely and relevant access** to the MH programs of the territorial health network of the EEPs that will participate in the project, thanks to the articulation of intersectoral networks that will be promoted.

## 3. Aim:

The team of researchers hopes to know the real possibilities of the application and effectiveness of an intervention that contemplates the training of teachers in SMI, in a hybrid modality, through a program co -constructed with the teachers participating in the present investigation, in order to to enhance their research and referral capacities to the Chilean public health system, to enhance access to timely and relevant intervention, with the support of a network of institutions, from different sectors, including: education, health, justice, among others. Others. Considering, in addition, that the return to school presence after the pandemic, will show the state of SM of children and adolescents in Chile who have been deprived of the sociability spaces provided by schools, restricted to the family space, which is not the norm in our culture. Therefore, we could expect the appearance of SM situations that require to be

addressed by specialized teams.

#### 4. Stake:

If you consent to your child's participation, you will be asked to complete the Strengths and Difficulties Questionnaire (SDQ) which screens for likely cases of mental and behavioral disorders in children ages 4-16 and that the head teacher of Your child can do it too. In addition, you will be required to provide information on whether the student is in mental health care.

Additional information: You will be informed via email or phone call, if the results of the instrument show a score of suspected mental health problem, and if you wish, this information will be delivered to the establishment's psychosocial team so that they can proceed with make a referral to the health network.

## 5. Costs and payments:

There will be no cost to you or your child to participate in this study. All activities are absolutely free, since FONIS and the University of Valparaíso cover all expenses associated with this study. Neither you nor your child will receive any financial compensation for their participation in the study. All activities associated with research will be carried out in the educational establishment.

#### 6. Profits:

It is expected that this project will report a benefit for the progress of skills in basic education teachers, specifically in early identification of SM difficulties that may arise in boys and girls with whom they have a daily relationship based on teaching work. contributing to generate timely and relevant access to health programs. Your child's participation in this study will not provide any additional direct benefits.

# 7. Risks:

We make it clear that there are no potential risks in this study, neither physical, nor emotional, nor of any kind for your child. On the other hand, the results would make it possible to have an intervention to improve SM in EEP boys and girls, with its initial evidence on effectiveness and feasibility indicators, for its possible scaling up to the national level. The application of the SDQ questionnaire to parents will be carried out by SM professionals. Therefore, a study that has a favorable risk/benefit balance is considered.

### 8. Confidentiality:

All information derived from your child's participation in this study will be kept strictly confidential, which includes access by researchers or research supervising agencies, by storing the documentation in locked cabinets, in offices of the School of Medicine of the University of Valparaíso. Likewise, the databases that will be used for statistical analysis will be built without including information that allows knowing the identity of the people who participated in the study (anonymous). In addition, any publication or scientific communication of the research results will be completely anonymous.

#### 9. Use and Publication of the findings

The results of this study will be disseminated through different public channels, either in the form of publications (scientific articles) or presentations (exhibition at conferences and congresses). In addition, we hope that the technology that we will evaluate through this research will be transferred to public services later.

#### 10. Bioethics Committee evaluation and contact:

This research has been evaluated and accepted by the Institutional Committee for Research Bioethics in Human Beings of the University of Valparaíso. If you require it, you can contact any of its members with its administrative secretary, Ms. Patricia Arancibia Pardo, on the phone +56 32-2507909, or through the institutional email cec.uv@uv.cl.

After having received and understood the information in this document and having been able to clarify all my doubts, I give my consent for my son/daughter to be given the qualities and difficulties questionnaire: SDQ

If you decide that the SDQ questionnaire will **NOT** be applied to your child, we ask you to sign this document

| Caregiver name: Investigator RUT: Date: | Researcher name: Eva Madrid Aris<br>Investigator RUT: 6.890.922-8<br>Date: |
|---|---|
| Firm: | Firm: |

Valparaiso, March 2023